CLINICAL TRIAL: NCT04827251
Title: Evaluation of the Effect of Espresso on Platelet Aggregability in Patients with Coronary Artery Disease
Brief Title: Effects of Espresso on Platelet Aggregability in Patients with Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Director of Coronary Care Unit, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SDC 4954/19/173
Record Dates: First submitted 2021-03-19; First posted 2021-04-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coffee; platelet aggregation; caffeine; aggregability
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coffee

STUDY DESIGN:
Intervention Model Description: This is a prospective, open label, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeinated coffee (Other): Patients will be instructed to abstain from caffeinated beverages during 22 days. After this period, they will consume caffeinated coffee during 28 days, followed by decaffeinated coffee during more 28 days.
  Interventions: Dietary Supplement: Coffee
- Decaffeinated coffee (Other): Patients will be instructed to abstain from caffeinated beverages during 22 days. After this period, they will consume decaffeinated coffee during 28 days, followed by caffeinated coffee during more 28 days.
  Interventions: Dietary Supplement: Coffee

INTERVENTIONS:
Dietary Supplement: Coffee — Participants will receive "Nespresso" coffee maker "Essenza" model. The coffee "Nespresso blend voluto" will be provided (caffeinated and decaffeinated). The patients will have to take four cups of espresso per day (three cups a day for patients aged 65 and over).

SUMMARY:
Discovered thousands of years ago, coffee is among the most consumed beverages in the world. The relationship between coffee and cardiovascular risk, more specifically coronary artery disease, is controversial. Platelet aggregation and its relationship with coffee is also controversial. The investigators propose this study to evaluate the relationship between coffee and platelet aggregability in patients with coronary artery disease.

DETAILED DESCRIPTION:
30 patients with coronary artery disease (proven by previous coronary angiography) will be selected at the Heart Institute (InCor USP) for the study. Patients will be instructed to abstain from caffeinated beverages during 22 days. After this period, one group will consume caffeinated coffee during 28 days, followed by decaffeinated coffee during more 28 days and another group will start with decaffeinated coffee followed by caffeinated. All participants will receive "Nespresso" coffee maker "Essenza" model. The coffee "Nespresso blend voluto" will be provided (caffeinated and decaffeinated). The patients will have to take four cups of espresso per day (three cups a day for patients aged 65 and over). The investigators will evaluate platelet aggregation by Multiplate® (ASPI, ADP and arachidonic acid) and by optical aggregometry (ADP and arachidonic acid).

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 years;
* Coronary artery disease documented by coronary angiography;
* Use of aspirin 100mg.

Exclusion Criteria:

* Serum creatinine dosage > 2.5 mg/dl;
* Hemoglobin <12 g/% for men and <11 g/% for women;
* Platelets <100,000 or >400,000/mm3;
* Leukocytosis >12,000/mm3;
* Fasting glycemia >126mg/dl;
* Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) with values above the upper limits of normality;
* Consumption of more than 30 grams of alcohol per day;
* Active smoking or ex-smoking for less than 2 years;
* Use of P2Y12 inhibitor;
* Ventricular dysfunction (left ventricular ejection fraction <45%).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation evaluated by Multiplate® ASPI | 8 weeks (±1)
  Compare the inhibition of platelet aggregation evaluated by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period).

SECONDARY OUTCOMES:
Platelet aggregation evaluated by Multiplate® ADP e Arachidonic acid | 4 week (±1)
  Compare the inhibition of platelet aggregation evaluated by Multiplate® ADP and Arachidonic acid after 4 weeks of caffeinated coffee consumption with platelet aggregability after 4 weeks of decaffeinated coffee consumption.
Platelet aggregation evaluated by Multiplate® ADP | 8 weeks (±1)
  Compare the inhibition of platelet aggregation evaluated by Multiplate® ADP after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period).
Platelet aggregation evaluated by optical aggregometry (ADP and arachidonic acid) 1 | 8 weeks (±1)
  Compare platelet aggregability by optical aggregometry (ADP and arachidonic acid) after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period).
Platelet aggregation evaluated by optical aggregometry (ADP and arachidonic acid) | 4 weeks (±1)
  Compare the inhibition of platelet aggregation evaluated by optical aggregometry (ADP and arachidonic acid) after 4 weeks of caffeinated coffee consumption with platelet aggregability after 4 weeks of decaffeinated coffee consumption.

OTHER OUTCOMES:
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: Elderly (≥65 years) and non-elderly | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: Elderly (≥65 years) and non-elderly
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: Feminine and masculine genders | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: Feminine and masculine genders
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: Renal dysfunction (Creatinine > 1.8mg/dl) and without renal dysfunction | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: Renal dysfunction (Creatinine > 1.8mg/dl) and without renal dysfunction
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: Obese (BMI≥30 Kg/m2) and non-obese | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: Obese (BMI≥30 Kg/m2) and non-obese
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: Glycemia >99mg/dl and no change in fasting glycemia | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: Glycemia >99mg/dl and no change in fasting glycemia
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: With of Beta-blocker and without | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: With of Beta-blocker and without
Compare platelet aggregation by Multiplate® ASPI in the following subgroup: With statin and without | 8 weeks (±1)
  Compare platelet aggregation by Multiplate® ASPI after 8 weeks of espresso consumption in relation to basal platelet aggregability (after coffee withdrawal period) in the following subgroup: With statin and without
Delta change of platelet aggregation and Fraction of immature platelets (PFI) | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Fraction of immature platelets (PFI)
Delta change of platelet aggregation and Small-LDL | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Small-LDL
Delta change of platelet aggregation and Fasting glycemia | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Fasting glycemia
Delta change of platelet aggregation and Glycated hemoglobin | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Glycated hemoglobin
Delta change of platelet aggregation and Lipid profile | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Lipid profile (total cholesterol, HDL [high-density lipoprotein], LDL [low-density lipoprotein], very low-density lipoprotein [VLDL] and triglycerides)
Delta change of platelet aggregation and Lipoprotein a | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Lipoprotein a - Lp(a)
Delta change of platelet aggregation and Sirtuins | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Sirtuins
Delta change of platelet aggregation and Advanced glycation final product (RAGE) receiver | 8 weeks (±1)
  Correlate the delta change of platelet aggregation of the basal in relation to 8 weeks of coffee use in relation to: Advanced glycation final product (RAGE) receiver

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adriana Farah. Coffee: Emerging Health Effects and Disease Prevention. Coffee Constituints. 2012. John Wiley & Sons, Inc. Published by Blackwell Publishing Ltd.
- [Background] Greenberg JA, Chow G, Ziegelstein RC. Caffeinated coffee consumption, cardiovascular disease, and heart valve disease in the elderly (from the Framingham Study). Am J Cardiol. 2008 Dec 1;102(11):1502-8. doi: 10.1016/j.amjcard.2008.07.046. Epub 2008 Sep 11. PMID 19026304
- [Background] Wu JN, Ho SC, Zhou C, Ling WH, Chen WQ, Wang CL, Chen YM. Coffee consumption and risk of coronary heart diseases: a meta-analysis of 21 prospective cohort studies. Int J Cardiol. 2009 Nov 12;137(3):216-25. doi: 10.1016/j.ijcard.2008.06.051. Epub 2008 Aug 15. PMID 18707777
- [Background] Lopez-Garcia E, van Dam RM, Willett WC, Rimm EB, Manson JE, Stampfer MJ, Rexrode KM, Hu FB. Coffee consumption and coronary heart disease in men and women: a prospective cohort study. Circulation. 2006 May 2;113(17):2045-53. doi: 10.1161/CIRCULATIONAHA.105.598664. Epub 2006 Apr 24. PMID 16636169
- [Background] Rosner SA, Akesson A, Stampfer MJ, Wolk A. Coffee consumption and risk of myocardial infarction among older Swedish women. Am J Epidemiol. 2007 Feb 1;165(3):288-93. doi: 10.1093/aje/kwk013. Epub 2006 Nov 16. PMID 17110637
- [Background] Happonen P, Voutilainen S, Salonen JT. Coffee drinking is dose-dependently related to the risk of acute coronary events in middle-aged men. J Nutr. 2004 Sep;134(9):2381-6. doi: 10.1093/jn/134.9.2381. PMID 15333732
- [Background] LaCroix AZ, Mead LA, Liang KY, Thomas CB, Pearson TA. Coffee consumption and the incidence of coronary heart disease. N Engl J Med. 1986 Oct 16;315(16):977-82. doi: 10.1056/NEJM198610163151601. PMID 3762618
- [Background] Andersen LF, Jacobs DR Jr, Carlsen MH, Blomhoff R. Consumption of coffee is associated with reduced risk of death attributed to inflammatory and cardiovascular diseases in the Iowa Women's Health Study. Am J Clin Nutr. 2006 May;83(5):1039-46. doi: 10.1093/ajcn/83.5.1039. PMID 16685044
- [Background] Greenberg JA, Dunbar CC, Schnoll R, Kokolis R, Kokolis S, Kassotis J. Caffeinated beverage intake and the risk of heart disease mortality in the elderly: a prospective analysis. Am J Clin Nutr. 2007 Feb;85(2):392-8. doi: 10.1093/ajcn/85.2.392. PMID 17284734
- [Background] Ding M, Bhupathiraju SN, Satija A, van Dam RM, Hu FB. Long-term coffee consumption and risk of cardiovascular disease: a systematic review and a dose-response meta-analysis of prospective cohort studies. Circulation. 2014 Feb 11;129(6):643-59. doi: 10.1161/CIRCULATIONAHA.113.005925. Epub 2013 Nov 7. PMID 24201300
- [Background] Cavalcante et al. Influência da Cafeína no Comportamento da Pressão Arterial e da Agregação Plaquetária. Arq Bras Cardiol, volume 75 (nº 2), 97-101, 2000
- [Background] Stefanello N, Spanevello RM, Passamonti S, Porciuncula L, Bonan CD, Olabiyi AA, Teixeira da Rocha JB, Assmann CE, Morsch VM, Schetinger MRC. Coffee, caffeine, chlorogenic acid, and the purinergic system. Food Chem Toxicol. 2019 Jan;123:298-313. doi: 10.1016/j.fct.2018.10.005. Epub 2018 Oct 3. PMID 30291944
- [Background] Olas B, Brys M. Effects of coffee, energy drinks and their components on hemostasis: The hypothetical mechanisms of their action. Food Chem Toxicol. 2019 May;127:31-41. doi: 10.1016/j.fct.2019.02.039. Epub 2019 Mar 4. PMID 30844438
- [Background] Natella F, Nardini M, Belelli F, Pignatelli P, Di Santo S, Ghiselli A, Violi F, Scaccini C. Effect of coffee drinking on platelets: inhibition of aggregation and phenols incorporation. Br J Nutr. 2008 Dec;100(6):1276-82. doi: 10.1017/S0007114508981459. Epub 2008 Apr 28. PMID 18439332
- [Background] Bydlowski SP, Yunker RL, Rymaszewski Z, Subbiah MT. Coffee extracts inhibit platelet aggregation in vivo and in vitro. Int J Vitam Nutr Res. 1987;57(2):217-23. PMID 3115908
- [Background] Bak AA, van Vliet HH, Grobbee DE. Coffee, caffeine and hemostasis: results from two randomized studies. Atherosclerosis. 1990 Aug;83(2-3):249-55. doi: 10.1016/0021-9150(90)90170-n. PMID 2146967
- [Background] Varani K, Portaluppi F, Gessi S, Merighi S, Ongini E, Belardinelli L, Borea PA. Dose and time effects of caffeine intake on human platelet adenosine A(2A) receptors : functional and biochemical aspects. Circulation. 2000 Jul 18;102(3):285-9. doi: 10.1161/01.cir.102.3.285. PMID 10899090
- [Background] Ammaturo V, Perricone C, Canazio A, Ripaldi M, Ruggiano A, Zuccarelli B, Monti M. Caffeine stimulates in vivo platelet reactivity. Acta Med Scand. 1988;224(3):245-7. doi: 10.1111/j.0954-6820.1988.tb19368.x. PMID 2977050
- [Background] Hattesen AL, Modrau IS, Nielsen DV, Hvas AM. The absorption of aspirin is reduced after coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2019 Mar;157(3):1059-1068. doi: 10.1016/j.jtcvs.2018.08.088. Epub 2018 Sep 27. PMID 30401532
- [Background] Diffenderfer MR, Schaefer EJ. The composition and metabolism of large and small LDL. Curr Opin Lipidol. 2014 Jun;25(3):221-6. doi: 10.1097/MOL.0000000000000067. PMID 24811298
- [Background] Dhand, N. K., & Khatkar, M. S. (2014). Statulator: An online statistical calculator. Sample Size Calculator for Comparing Two Paired Means. Accessed 7 May 2019 at http://statulator.com/SampleSize/ss2PM.html
- [Background] Michan S, Sinclair D. Sirtuins in mammals: insights into their biological function. Biochem J. 2007 May 15;404(1):1-13. doi: 10.1042/BJ20070140. PMID 17447894
- [Background] Hofmann MA, Drury S, Fu C, Qu W, Taguchi A, Lu Y, Avila C, Kambham N, Bierhaus A, Nawroth P, Neurath MF, Slattery T, Beach D, McClary J, Nagashima M, Morser J, Stern D, Schmidt AM. RAGE mediates a novel proinflammatory axis: a central cell surface receptor for S100/calgranulin polypeptides. Cell. 1999 Jun 25;97(7):889-901. doi: 10.1016/s0092-8674(00)80801-6. PMID 10399917
- [Background] Hudson BI, Carter AM, Harja E, Kalea AZ, Arriero M, Yang H, Grant PJ, Schmidt AM. Identification, classification, and expression of RAGE gene splice variants. FASEB J. 2008 May;22(5):1572-80. doi: 10.1096/fj.07-9909com. Epub 2007 Dec 18. PMID 18089847